CLINICAL TRIAL: NCT05668767
Title: Multi-centered, Single-arm, Phase II Study on Surufatinib in Combination of Durvalumab and Etoposide and Carboplatin/Cisplatin in the Firstly-line Treatment of Extensive-stage Small-cell Lung Cancer
Brief Title: Surufatinib in Combination of Durvalumab and EP/EC in the Firstly-line Treatment of ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-N1-SCLC107
Record Dates: First submitted 2022-12-20; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Single-arm Surufatinib Durvalumab EP/EC
  Interventions: Drug: Surufatinib Durvalizumab EP/EC

INTERVENTIONS:
Drug: Surufatinib Durvalizumab EP/EC — Etoposide: total 100 mg/m2, once a day, continuous intravenous drip for more than 3 hours, days 1 to 3, q3w Cisplatin: total 75 mg/m2, once a day, continuous intravenous drip for more than 3 hours, days 1 to 3, q3w; or Carboplatin: AUC 5-6, intravenous infusion, administered on day 1 of each treatment cycle, q3w
  Other Names: HMPL-012

SUMMARY:
Though great progress has been made in the treatment of SCLC in recent years, only two PD-L1 therapies are currently approved, treatment options are limited, and patient survival remains to be further improved. The current study aims to investigate the efficacy and safety of surufatinib combined with durvalumab combined with EP/EC regimen in first-line treatment of patients with extensive-stage SCLC, and to further explore the predictive biomarkers of this treatment combination.

DETAILED DESCRIPTION:
BACKGROUND: Small-cell lung cancer (SCLC) is an aggressive neuroendocrine tumor derived from bronchial epithelial cells, accounting for about 13-15% of all lung cancers. It has a rapid doubling time and high growth fraction, and tends to metastasize widely early in the course of the disease, resulting in 95% mortality. It is the most lethal subtype of lung cancer.

Platinum-based chemotherapy is the first-line standard treatment for localized and extensive SCLC, with platinum combined with etoposide as the preferred regimen. However, chemotherapy options are limited and there remains a great unmet need for efficacy.

In recent years, with the development of immunotherapy, chemotherapy combined with immunization has also become the treatment option for treatment-naïve patients, and PD-L1 inhibitor combined with chemotherapy first-line treatment has become a guideline class 1A recommendation; there is a significant benefit in OS compared with chemotherapy: in the IMpower 133 study, atezolizumab combined with EP regimen resulted in an OS of 12.3 months; in the CASPIAN study, Durvalumab combined with EP/EC regimen resulted in an OS of 13 months.

An increasing number of targeted therapeutics have also been newly explored in the field of SCLC. In first-line treatment, PFS reached 9.6 months, OS reached 13.87 months, and ORR reached 77.8% with anlotinib in combination with EP/EC regimen.

Though great progress has been made in the treatment of SCLC in recent years, only two PD-L1 therapies are currently approved, treatment options are limited, and patient survival remains to be further improved. The current study aims to investigate the efficacy and safety of surufatinib combined with durvalumab combined with EP/EC regimen in first-line treatment of patients with extensive-stage SCLC, and to further explore the predictive biomarkers of this treatment combination.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. pathohistologically or cytologically confirmed small cell lung cancer with measurable lesions (RECIST 1.1, see Appendix 2);
3. no previous systemic anti-tumor therapy;
4. ECOG 0 or 1 (see Appendix 1);
5. expected survival ≥ 12 weeks;
6. at least one measurable lesion (RECIST 1.1 criteria);
7. basically normal major organ and bone marrow function: a) blood routine: white blood cells ≥ 4.0 x 109/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 90 g/L; b) international normalized ratio (INR) ≤ 1.5 × upper limit of normal (ULN), and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; c) liver function: total bilirubin ≤ 1.5 x ULN; in the absence of liver metastasis, ALT/AST/ALP ≤ 2.5 x ULN; in the presence of liver metastases,ALT/AST/ALP ≤ 5 x ULN; d) renal function: serum creatinine ≤ 1.5 x ULN, and creatinine clearance (CCr) 60 mL/min (see Appendix 6); e) normal cardiac function, left ventricular ejection fraction (LVEF) ≥ 50% by two-dimensional echocardiography.
8. fully understand the study, voluntarily participate, and sign the informed consent form.
9. male or female patients of childbearing potential voluntarily use effective contraceptive methods during the study and within 6 months of the last study medication, such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives, intrauterine devices, etc.All female patients will be considered to be of childbearing potential unless they are naturally postmenopausal, have undergone artificial menopause, or have undergone sterilization (eg, hysterectomy, bilateral adnexectomy, or radiation ovarian irradiation).

Exclusion Criteria:

1. previously received systemic anti-tumor therapy for small cell lung cancer;
2. tumors showing significant cavities or necrosis on imaging (CT or MRI)
3. patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination suggesting brain or leptomeningeal lesions) (patients with brain metastases within 28 days before the completion of randomized treatment and symptoms from stable enrollment, but brain MRI examination is required, and CT or intravenous angiography confirms no symptoms of cerebral hemorrhage);
4. patients who are participating in other clinical studies within 4 weeks after the end of previous clinical studies (except non-interventional studies);
5. Patients who have received chemotherapy, radiotherapy or other investigational anticancer therapy (except bisphosphonates) within 4 weeks prior to the first dose of this study. Patients who have previously received local radiotherapy are eligible if they meet the following criteria: end of radiotherapy more than 4 weeks from the start of this study (brain radiotherapy more than 2 weeks); in addition, the target lesions selected for this study are not in the radiotherapy area, or if the target lesions are within the radiotherapy area, but progression has been confirmed;
6. Other types of malignancy within 5 years or present;
7. patients with active, known, or suspected autoimmune diseases, including allogeneic organ transplantation, history of allogeneic hematopoietic stem cell transplantation, history of HIV-positive or history of acquired immunodeficiency syndrome (AIDS);
8. active or previously documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis);
9. non-remitting toxicity from previous treatment, more than CTC AE (4.0) grade 1, excluding alopecia;
10. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or receiving thrombolytic and anticoagulant therapy, clinically significant hemoptysis (hemoptysis more than half a tablespoon daily; or clinically significant bleeding symptoms or bleeding tendency within 4 weeks before grouping, such as gastrointestinal bleeding, hemorrhagic gastric ulcer (including gastrointestinal perforation and/or fistula, but gastrointestinal perforation or fistula has been surgically removed, admission is allowed), baseline fecal occult blood + + or more, unhealed wounds, ulcers or fractures;
11. urine routine showed urine protein ≥ + +, or urine protein ≥ 1.0 g within 24 hours;
12. Uncontrolled hypertension (SBP ≥ 160 mmHg and DBP ≥ 100 mmHg despite optimal medical therapy);
13. Patients with severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia; according to NYHA criteria, grade III-IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) < 50% by echocardiography;
14. Patients with NCI-CTCAE grade II or higher peripheral neuropathy, except due to trauma;
15. Interstitial lung disease, uncontrolled moderate to large serous effusion (including pleural effusion, ascites, and pericardial effusion) after pumping therapy, exacerbation of chronic obstructive pulmonary disease requiring intravenous antibiotics within 28 days, active pulmonary infection, and/or acute bacterial or fungal respiratory disease;
16. There are factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction;
17. Venous thromboembolic events such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis, pulmonary embolism within 6 months prior to enrollment;
18. Has received a live or attenuated vaccine within 30 days prior to the first dose of dulizumab, or plans to receive a live or attenuated vaccine during the study;
19. Known history of severe hypersensitivity to other monoclonal antibodies;
20. Known history of psychotropic drug abuse, alcohol abuse, or drug abuse;
21. Active hepatitis uncontrolled after treatment (hepatitis B: HBsAg positive and HBV DNA more than 1 x 10 ^ 4 copies/ml; hepatitis C: HCV RNA positive and abnormal liver function); combined hepatitis B and C infection;
22. Have other serious diseases that, in the opinion of the investigator, jeopardize the patient 's safety or affect the patient' s completion of the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival(PFS) | up to 24 months
  assessed by the investigator as per the Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Overall survival | About 18 months
  Overall survival (OS)
Objective response rate | About 18 months
  Objective response rate (ORR) assessed per RECIST v1.1
Disease control rate | About 18 months
  Disease control rate (DCR) assessed per RECIST v1.1
Quality of Life | About 18 months
  EORCT-QLQ-LC13 Scale
Incidence of adverse events | From Baseline to primary completion date, about 18 months
  The incidence of adverse events of all grades

IPD SHARING:
Plan to Share IPD: No